CLINICAL TRIAL: NCT00661921
Title: A Mutiple Dose, Randomized, Double-blind, Placebo-controlled Study of Subcutaneous AMG 108 in Patients With Type 2 Diabetes Mellitus
Brief Title: A Randomized Double Blind, Placebo Controlled Trial With AMG 108 in Patients With Type 2 Diabetes Mellitus
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Program Development discontinued
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20070212
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; AMG 108; HbA1C; glucose; metformin; sulfonylurea; IL-1 Inhibitor; biologic; subcutaneous injection
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — AMG 108

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 40 mg AMG 108 Q2W (Active Comparator)
  Interventions: Biological: AMG 108
- 150 mg AMG 108 Q2W (Active Comparator)
  Interventions: Biological: AMG 108
- 75 mg AMG 108 Q2W (Active Comparator)
  Interventions: Biological: AMG 108
- Placebo Q2W (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AMG 108 — IL-1 inhibitor, subcutaneous injection given every 2 weeks for the duration of the trial. Doses include 150 mg, 75mg, and 40 mg.
  Arms: 150 mg AMG 108 Q2W; 40 mg AMG 108 Q2W; 75 mg AMG 108 Q2W
Biological: Placebo — AMG 108 volume matching placebo
  Arms: Placebo Q2W

SUMMARY:
The purpose of this study is to investigate the effects of blocking IL-1 signaling with AMG 108 in type 2 diabetes mellitus patients on glycemic control, as measured by change in HbA1c from baseline to end of treatment (EOT).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM ≥ 3 months at time of randomization
* HbA1c of 7.0 - 9.5% (inclusive) at screening
* ≥ 18 years of age at the time of randomization
* BMI ≥ 25 kg/m2 and ≤ 45 kg/m2 at screening, and, per patient self-report, following their regular weight maintenance or reduction diet for the management of diabetes for at least 4 weeks prior to randomization
* Fasting plasma glucose ≤ 240 mg/dL (13.3 mmol/L) at each of 2 determinations during screening (samples taken at least 1 day apart)
* No new therapy for the treatment of elevated blood pressure or dyslipidemia, use of any weight loss medication (over the counter or prescription), or initiation of a prescribed weight management or exercise program within 4 weeks before randomization
* Subject is able and willing to comply with the study's visit requirement

Exclusion Criteria:

* History of type 1 insulin-dependent diabetes
* Significant signs and symptoms of uncontrolled hyperglycemia (ie, polyuria, polydypsia, polyphagia), in the opinion of the investigator
* History of significant weight gain or loss (+/- 5%) during the 4 weeks before randomization
* Triglycerides ≥ 400 mg/dL (4.5 mmol/L) and/or total cholesterol ≥340 mg/dL (8.7 mmol/L) at screening
* Currently receiving or received within 60 days prior to screening any anti-diabetic pharmaceutical therapy (eg, insulin) other than metformin and/or sulfonylurea. If receiving metformin or sulfonylurea, doses must be stable for ≥ 60 days.
* Uncontrolled hypertension defined as diastolic pressure > 95 mmHg and/or systolic > 170 mmHg during screening
* Hepatic function test (alanine aminotranferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, total bilirubin) results at screening > 2 times the upper limit of normal for the central laboratory
* White blood cell count < 3000 / μL, absolute neutrophil count (ANC) of < 2500 / μL, or platelet count of < 125,000 / μL at screening
* Any significant inflammatory, rheumatologic, or systemic autoimmune disease in the opinion of the investigator
* Evidence of active infection, recent infection, or chronic infection, requiring treatment with anti-infectives, hospitalization or IV antibiotics within 4 weeks prior to randomization
* Active or latent Mycobacterium tuberculosis infection as defined by known positive PPD or chest x-ray findings and failure to complete treatment with appropriate chemoprophylaxis, or exposure to a person with active tuberculosis within 6 months prior to randomization
* Existence of non-healing wounds or ulcers
* Known to be positive for hepatitis B surface antigen (HbsAg), hepatitis C virus (HCV) or human immunodeficiency virus (HIV)
* Estimated GFR (eGFR) at screening < 30 mL/min as calculated via the MDRD equation (Modification of Diet in Renal Disease study group)
* Clinical evidence of current malignancy, with the following exceptions: basal or squamous cell carcinoma of the skin, cervical intraepithelial neoplasia, prostate cancer (if stable localized disease, with life expectancy of > 3 years); or receiving or has received chemotherapy and/or radiation therapy for treatment of a malignancy within 6 months prior to randomization
* Clinically significant cardiovascular disease (eg, heart failure of New York Heart Association [NYHA] class 3 or 4), hematological abnormality, asthma, or chronic obstructive pulmonary disease (eg, requiring oral or IV steroids), in the opinion of the investigator
* Receipt of any biologic or immunosuppressive therapy (experimental or commercial), including anakinra (Kineret®) or any tumor necrosis factor (TNF) blocking agents (eg, etanercept and infliximab), or live vaccines, within 3 months of randomization
* Previously received AMG 108
* Subject is evidently pregnant (eg, positive human chorionic gonadotropin [HCG] test), is breast feeding, or is of child-bearing potential and not using adequate contraceptive precautions, as determined by the investigator
* Subject currently is enrolled in or has not yet completed at least 30 days since ending other investigational device or drug study(s), or subject is receiving other investigational agent(s)
* Subject has any kind of condition (eg, psychiatric illness) or situation that, in the investigator's opinion, compromises the ability of the subject to give written informed consent, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2009-06 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HbA1c at week 14 (end of treatment) | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com